CLINICAL TRIAL: NCT01531777
Title: A Random, Open, Dose Finding and Pharmacokinetics/Pharmacodynamics(PK/PD) Phase II Study of Apatinib Tablets in the Treatment of Advanced Colorectal Cancer
Brief Title: Dose Finding and Pharmacokinetics/Pharmacodynamics Study of Apatinib in the Treatment of Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APTN-II-CRC
Record Dates: First submitted 2012-02-07; First posted 2012-02-13 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer
Keywords: Advanced Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apatinib 500mg (Experimental): 500mg,p.o.,qd
  Interventions: Drug: Apatinib
- Apatinib 750mg (Experimental): 750mg,p.o.,qd
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: Apatinib — 500 mg,p.o.,qd, until disease progression or intolerable toxicity or patients withdrawal of consent.
  Arms: Apatinib 500mg
Drug: apatinib — 750 mg,p.o.,qd, until disease progression or intolerable toxicity or patients withdrawal of consent.
  Arms: Apatinib 750mg

SUMMARY:
RATIONALE:

Apatinib is a tyrosin-inhibitor agent targeting at vascular endothelial growth factor receptor (VEGFR), and it's anti-angiogenesis effect has been viewed in preclinical tests. The investigators' phase I study has shown that the drug's toxicity is manageable.

PURPOSE:

1. Studying how well Apatinib works in treating patients.
2. Finding the efficacy and safety of 500 mg or 750mg Apatinib.
3. Pharmacokinetics/Pharmacodynamics(PK/PD).
4. Exploring new outcome measures of antiangiogenic drugs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age
* Histological confirmed advanced or metastatic colorectal Cancer，at least one measurable lesion, larger than 10 mm in diameter by spiral CT scan(scanning layer ≤ 5 mm )
* Have failed for ≥ 2 lines of chemotherapy
* Life expectancy of more than 3 months
* ECOG performance scale ≤ 1
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin More than 4 weeks for operation, radiotherapy or cytotoxic agents
* Adequate hepatic, renal, heart, and hematologic functions (platelets > 80 × 10E+9/L, neutrophil > 1.5 × 10E+9/L, serum creatinine ≤ 1×upper limit of normal(ULN), bilirubin < 1.25 ULN, and serum transaminase ≤ 2.5× ULN)
* Child bearing potential, a negative urine or serum pregnancy test result before initiating apatinib, must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article.
* Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg despite using single medical therapy, more than class I (NCI CTCAE 3.0 ) myocardial ischemia, arrhythmia(including QTcF:male ≥ 450 ms, female ≥ 470 ms), or cardiac insufficiency myocardial ischemia, arrhythmia, or cardiac insufficiency
* Before or at the same time any, second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Any factors that influence the usage of oral administration Evidence of CNS metastasis
* URT: urine protein ≥ (++)and > 1.0 g of 24 h
* PT, APTT, TT, Fbg abnormal, having hemorrhagic tendency (eg. active peptic ulcer disease) or receiving the therapy of thrombolysis or anticoagulation
* Abuse of drugs
* Certain possibility of gastric or intestine hemorrhage
* Less than 4 weeks from the last clinical trial
* Viral hepatitis type B or type C
* Prior VEGFR inhibitor treatment
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | 12 weeks

SECONDARY OUTCOMES:
DCR (Disease Control Rate) | 12 weeks after treatment
PFS | 3 years
OS (Overall Survival) | 3 years
QoL (Quality of Life) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University cancer hospital, Shanghai, Shanghai Municipality, China